CLINICAL TRIAL: NCT00591162
Title: Bone Disease in Severely Burned Children
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: terminated due to PI lab/duties affected by natural disaster.
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 92-304
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-06

CONDITIONS: Burn
Keywords: Bone, Dexa, Parathyroid, Diuretic, Tetracycline
MeSH Terms: conditions — Burns | interventions — Tetracycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Active Comparator): Compare bone density of severly burned children to normal non-burned population
  Interventions: Drug: Tetracycline; Radiation: Duel Energy X-Ray Absorptiometry (DEXA); Procedure: Bone Biopsy

INTERVENTIONS:
Drug: Tetracycline — Two courses of IV Tetracycline(10mg./kg./day for two days)separated by a two week interval.
Radiation: Duel Energy X-Ray Absorptiometry (DEXA) — DEXA before discharge from acute admission and again one year post burn.
  Other Names: Duel Energy X-Ray Absorptiometry
Procedure: Bone Biopsy — Bone biopsy to be taken in the operation room at the last skin grafting operation at the site of the iliac crest. A second bone biopsy will be taken one year later post discharge from the acute admission.

SUMMARY:
Bone metabolism is adversely affected by severe burns in children for a period of time.

DETAILED DESCRIPTION:
More closely monitored biochemical and radiologic parameters of bone and mineral metabolism will increase the likelihood of earlier detection of abnormalities and possible therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

* Children age 5-18 years old with at least 40% or more of their body burned.

Exclusion Criteria:

* Anyone with a burn covering less than 40% of the body or whose burn covers the front of both hipbones.
* Anyone younger than 5 years old, anyone with a history of cancer or other metabolic disease process, or anyone who is pregnant or has an allergy to Tetracycline will also be excluded.
* Anyone who has participated in an investigational drug trial within the past 60 days from date of admission will be excluded from this study.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 254 (Actual)
Dates: Start 1992-10; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Determine Bone Health(bone growth,strength,and content) in burn injured patients. | Admission to Burn Unit up to eighteen years old.

CONTACTS AND LOCATIONS:
Overall Officials: Klein Gordon, M.D., Principal Investigator — U.T.M.B.
Locations (1):
- U.T.M.B., Galveston, Texas, United States